CLINICAL TRIAL: NCT01204528
Title: Diastolic Dysfunction, Microcirculation Disturbance, Sympathetic Activation and Inflammation in Moderate Kidney Failure and in Diabetic Nephropathy: Disease Modification With Vitamin-D Receptor Activation. A Double-blind, Placebo-controlled, Randomised Trial - the SOLID Trial
Brief Title: Vitamin-D Receptor Activation (VDRA) in Chronic Kidney Disease
Acronym: SOLID
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Jonas Spaak, MD, PhD, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VDRA
Record Dates: First submitted 2010-04-27; First posted 2010-09-17 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Kidney Disease
Keywords: Dysfunction in CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Paricalcitol 2 microgram/d (Active Comparator)
  Interventions: Drug: Zemplar
- Paricalcitol 1 microgram/d (Active Comparator)
  Interventions: Drug: Zemplar
- Placebo (Placebo Comparator)
  Interventions: Drug: Zemplar

INTERVENTIONS:
Drug: Zemplar — Vitamin D receptor activator (VDRA)

SUMMARY:
To investigate whether treatment with a vitamin-D receptor activator is able to improve important markers of cardiovascular risk.

DETAILED DESCRIPTION:
Main question:

May 12 weeks of VDRA treatment reduce the pathological sympathetic overactivation associated with moderate kidney disease?

Secondary questions aim to thrown light on how VDRAs can reduce albuminuria and CRP, i.e. does VDRA treatment improve (prespecified statistical analyses):

A) diastolic dysfunction? B) capillary microcirculation, and whether ameliorated disturbances relate to improved diastolic dysfunction? C) endothelial dysfunction and arterial stiffness? D) inflammatory activation? E) platelet function and haemostasis? F) levels of antibacterial peptides? G) levels of IGFBP-1 and adiponectin?

Overall design The study is designed as a double-blind, randomised, placebo-controlled trial involving two groups (n=72) of patients: 1) chronic kidney failure (CKD, eGFR 15-59 mL/m2) and 2) chronic kidney failure and concomitant diabetes mellitus (CKD+DM).

It will start with a two-week placebo run-in, followed by randomisation to:

1. Zemplar 1 μg (taken as 1 x 1 μg capsule and one placebo capsule),
2. Zemplar 2 μg (taken as 2 x 1 μg capsules) and
3. placebo (taken as two placebo capsules).

ELIGIBILITY:
Inclusion Criteria:

eGFR 15-59 ml/m2

Exclusion Criteria:

Current vitamin D treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-09; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
A significant reduction in muscle sympathetic nerve activity (MSNA) measured by means of microneurography. | Measured after 12 weeks treatment.
  Sympathetic activation is closely related to severity and progression of cardiovascular diseases, and renovascular dysfunction. We will directly measure sympathetic activation using microneurography (muscle sympathetic nerve activity; MSNA), expressed as bursts/minute and bursts/100 RR-interval. As this is a physiological study, the primary outcome will constitute a significant reduction in MSNA.

SECONDARY OUTCOMES:
Microcirculatory function measured by laser doppler methods. | Measured after 12 weeks treatment.
  Assessed by skin laser-doppler methodology, and directly by nailfold capillaroscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institute at Danderyd University Hospital, Danderyd, Stockholm County, Sweden

REFERENCES:
- [Derived] Lundwall K, Mortberg J, Mobarrez F, Jacobson SH, Jorneskog G, Spaak J. Changes in microparticle profiles by vitamin D receptor activation in chronic kidney disease - a randomized trial. BMC Nephrol. 2019 Aug 1;20(1):290. doi: 10.1186/s12882-019-1445-4. PMID 31370809
- [Derived] Mansouri L, Lundwall K, Moshfegh A, Jacobson SH, Lundahl J, Spaak J. Vitamin D receptor activation reduces inflammatory cytokines and plasma MicroRNAs in moderate chronic kidney disease - a randomized trial. BMC Nephrol. 2017 May 16;18(1):161. doi: 10.1186/s12882-017-0576-8. PMID 28511692
- [Derived] Lundwall K, Jorneskog G, Jacobson SH, Spaak J. Paricalcitol, Microvascular and Endothelial Function in Non-Diabetic Chronic Kidney Disease: A Randomized Trial. Am J Nephrol. 2015;42(4):265-73. doi: 10.1159/000441364. Epub 2015 Oct 24. PMID 26496210